CLINICAL TRIAL: NCT04572100
Title: Pilot Study of Induction Chemotherapy Followed by Risk and Response-Stratified Treatment for Locoregional HPV Associated Oropharyngeal Cancer
Brief Title: Pilot Study of Chemotherapy for HPV-Associated Oropharyngeal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB20-0713
Record Dates: First submitted 2020-09-17; First posted 2020-10-01 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma
Keywords: Oropharyngeal squamous cell carcinoma; head and neck cancer; HPV; human papillomavirus; OPSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Radiotherapy; Drug Therapy; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A - Low Risk (Experimental): Participants who have low-risk cancer and significant reduction (greater than 50%) in tumor size following induction therapy will be assigned to this group.
  Interventions: Other: Transoral Robotic Surgery (TORS) or Radiotherapy
- Group B - Intermediate Risk (Experimental): Participants who have low-risk cancer and intermediate reduction (30-50%) in tumor size or high-risk cancer with significant reduction (greater than or equal to 50%) in tumor size following induction therapy will be assigned to this group.
  Interventions: Other: Chemotherapy and Low-Dose Radiotherapy
- Group C - High-Risk (Experimental): Participants who have high-risk cancer and less than a 50% reduction in their tumor size following induction therapy will be assigned to this group.
  Interventions: Other: Chemotherapy and High-Dose Radiotherapy
- Induction Therapy (Carboplatin and Paclitaxel) (Experimental): All study participants will be assigned to this group to first receive induction therapy using a combination of carboplatin and paclitaxel. Participant response to this phase of therapy will determine which group (low-risk, intermediate risk or high-risk) the participant will be in.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Other: Transoral Robotic Surgery (TORS) or Radiotherapy — Participants assigned to this group will receive transoral robotic surgery (TORs) or radiotherapy. Radiotherapy is given once a day for 5 weeks. A percentage of subjects who undergo surgery may need further radiotherapy with or without chemotherapy based on the results of the surgery. TORs is surgery in which a robot with arms is used to remove cancer from hard-to-reach areas of the mouth and throat.
  Arms: Group A - Low Risk
Other: Chemotherapy and Low-Dose Radiotherapy — Participants assigned to this group will receive 5 weeks of chemotherapy combined with low- dose radiotherapy.
  Arms: Group B - Intermediate Risk
Other: Chemotherapy and High-Dose Radiotherapy — Participants assigned to this group will receive 7 weeks of chemotherapy combined with high- dose radiotherapy.
  Arms: Group C - High-Risk
Drug: Paclitaxel — This drug will be combined with carboplatin during induction therapy for 9 weeks.
  Other Names: Taxol
  Arms: Induction Therapy (Carboplatin and Paclitaxel)
Drug: Carboplatin — This drug will be combined with paclitaxel during induction therapy for 9 weeks.
  Other Names: Paraplatin
  Arms: Induction Therapy (Carboplatin and Paclitaxel)

SUMMARY:
Doctors leading this study will give blood tests to head and neck cancer participants during the beginning of chemotherapy treatment (also known as induction therapy) to see if these blood tests can help predict tumor shrinkage after therapy and reduce the amount of additional radiotherapy or chemotherapy treatment the participant may need. This study will also examine ways to reduce overall side effects of treatment using robotic surgery, chemotherapy and radiotherapy, or radiotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have clinically confirmed Human papillomavirus(HPV)-positive head and neck squamous cell cancer of the back of the mouth/throat (oropharynx). Confirmed HPV-positive disease of other subsites are uncommon but also eligible.
2. HPV testing must be compliant with the following criteria:

   1. P16INK4a immunohistochemistry (p16 IHC) positivity is sufficient to enroll and initiate treatment (p16 IHC interpretation to follow guidelines by Jordan and Lingen et al72).
   2. p16 IHC positivity is to be validated using an HPV Polymerase chain reaction (PCR - a type of DNA copying method).
   3. HPV PCR must demonstrate HPV16 or HPV18 subtype
3. Availability of greater than 10 unstained 5 micron slides (to be provided to HTRC at the University of Chicago). Patients who cannot fulfill this requirement will need to undergo a new biopsy prior to enrollment on study.
4. Participants must be at least 18 years old.
5. Participants with American Joint Committee on Cancer (AJCC) (8th edition, 2018) N1 (>=3cm), N2-N3 nodal disease or T3-T4 primary tumor.
6. Measurable disease (either primary site or nodal disease) according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 criteria.
7. No previous radiation or chemotherapy for a head and neck cancer.
8. No complete surgical resection for a head and neck cancer within 8 weeks of enrollment (although lymph node biopsy including excision of an individual node with presence of residual nodal disease, or surgical biopsy/excision of the tumor with residual measurable disease is acceptable.) No surgical procedures or biopsies will occur after baseline scans are performed and measurable lesions are identified.
9. Eastern Cooperate Oncology Group performance status 0-1
10. Normal organ function clinically confirmed by medical records.
11. Participants must sign a study-specific informed consent form prior to study entry. Participants should have the ability to understand and the willingness to sign a written informed consent document.
12. Women of childbearing potential must have a negative serum or urine pregnancy test within 24 hours prior to the start of study drug.
13. Women must not be breastfeeding.
14. Women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment.
15. Men who are sexually active with women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s).

Exclusion Criteria:

1. Any sign of metastatic disease (M1 disease).
2. Non-HPV16/18 subtype
3. Unidentifiable primary site of cancer.
4. Other medical illnesses that may impair the participant's ability to receive therapy or limit survival. This includes but is not limited to ongoing or active infection, immunodeficiency, symptomatic congestive heart failure, pulmonary dysfunction, cardiomyopathy, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance. Patients with clinically stable and/or chronically managed medical illnesses that are not symptomatic and/or are not expected to impact treatment on protocol are still eligible (conditions to be reviewed by the PI to confirm eligibility)
5. Prior surgical therapy other than incisional/excisional biopsy or organ-sparing procedures such as debulking of airway-compromising tumors. Residual measurable tumor is required for enrollment as discussed above.
6. Patients receiving other investigational agents.
7. Prior systemic anti-cancer treatment within the last 8 weeks.
8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer or any tumors that are not likely to influence life expectancy in the subsequent 3 years without active treatment.
9. Has known history of, or any evidence of active, non-infectious pneumonitis.
10. Has a history of HIV.
11. Has known active Hepatitis B or hepatitis C. If eradicated, patient is eligible.
12. Has received a live vaccine within 28 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of collection of serial HPV-DNA blood samples in patients undergoing treatment for Oropharyngeal Squamous Cell Carcinoma | 16 weeks
  To determine if it is possible (feasibility) to measure HPV-DNA using blood tests among participants undergoing induction chemotherapy followed by a second round of response-based therapy for their HPV-associated cancer. This feasibility will be determined by measuring the proportion of patients who complete chemotherapy treatment and HPV-DNA assessments.
Relationship Between HPV-DNA Found in Participant's Blood and Participant Response to Chemotherapy | 16 weeks
  To evaluate the relationship (aka correlation) between the amount of HPV-DNA found in a participant's plasma/blood and the participant's response to induction chemotherapy based on how their tumor responds to treatment.

SECONDARY OUTCOMES:
Changes in Blood Containing HPV-DNA During Response-Based Therapy | 16 weeks
  To evaluate changes in blood containing HPV-DNA during a second round of chemotherapy (known as response-based chemo-radiotherapy) that will be based on how the participant responded to their first/induction phase of chemotherapy treatment. This outcome will be measured by checking quantitative HPV DNA in plasma with each cycle of induction chemotherapy, weekly during radiation treatment, and following completion of radiation at set time points within the study.
Side Effects of Cisplatin-Based Chemotherapy Treatment | 16 weeks
  To evaluate the side effects of weekly cisplatin-based treatment in participants receiving chemotherapy followed by a second round of response-based therapy for their HPV-associated cancer.
Tumor Response Among Participants Undergoing Transoral Robotic Surgery | 20 weeks
  To determine how participant's tumor/cancer responds when they are undergoing Transoral Robotic Surgery (TORS) following induction chemotherapy. TORs is surgery in which a robot with arms is used to remove cancer from hard-to-reach areas of the mouth and throat. Data about how patients' tumors respond in this study will be compared to similar data from a previous study.
Time to Disease Recurrence | 5 years
  Length of time participants remain without evidence of disease.
Overall Survival | 5 years
  Length of time until participant death.
Locoregional Control | 5 years
  Number of participants who experience local control of their primary tumors after treatment.
Distant Control | 5 years
  Number of participants who experience control of metastatic disease (distant tumors) after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ari Rosenberg, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Rosenberg AJ, Izumchenko E, Pearson A, Gooi Z, Blair E, Karrison T, Juloori A, Ginat D, Cipriani N, Lingen M, Sloane H, Edelstein DL, Keyser K, Fredebohm J, Holtrup F, Jones FS, Haraf D, Agrawal N, Vokes EE. Prospective study evaluating dynamic changes of cell-free HPV DNA in locoregional viral-associated oropharyngeal cancer treated with induction chemotherapy and response-adaptive treatment. BMC Cancer. 2022 Jan 3;22(1):17. doi: 10.1186/s12885-021-09146-z. PMID 34980038